CLINICAL TRIAL: NCT00166127
Title: Pharmacokinetics and Pharmacodynamics of Levosimendan During Cardiac Surgery
Brief Title: Study of Blood Concentrations and Physiologic Effects of Levosimendan Given During Heart Surgery
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Unable to renegotiate an expired contract w/sponsor providing study med
Sponsor: Emory University (Other)
Collaborators: Abbott (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0984-2003; 6-38989
Record Dates: First submitted 2005-09-12; First posted 2005-09-14 (Estimated); Last update posted 2013-11-15 (Estimated); Status verified 2013-11

CONDITIONS: Heart Failure
Keywords: heart failure; cardiac surgery; pharmacokinetics; pharmacodynamics
MeSH Terms: conditions — Heart Failure | interventions — Simendan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Levosimendan

SUMMARY:
The purpose of this study protocol is to evaluate the blood concentrations of levosimendan when administered at different doses clinically employed during cardiopulmonary bypass or cardiac manipulation during off pump surgery in patients who require the drug for inotropic support (improved heart function) and the associated hemodynamic variables (vital signs). Levosimendan is one of the first agents in a new class of drugs used to treat heart failure and works via a unique mechanism called calcium sensitization, that makes the heart beat more efficiently. Levosimendan also has unique effects on the blood vessels, as well as causing relaxation, an important therapeutic approach of heart failure therapy.

DETAILED DESCRIPTION:
This is a non-randomized trial, and the patients will be assigned to one of three dose groups following cardiopulmonary bypass or prior to manipulation of the heart in the off pump group. A total of 30 patients will be enrolled into this study, 20 off-pump and 10 subjects on pump. Levosimendan is approved in Europe for the treatment of decompensated heart failure. It improved cardiac function without increasing energy demands. The subject's enrollment ends at Day 7 or day of discharge, whichever comes first.

ELIGIBILITY:
Inclusion Criteria:

* At least 21 years of age
* Less than 80 years of age
* ASA Class III-IV
* Scheduled for elective cardiac surgery
* Signed informed consent
* History of heart failure, and/or left ventricular ejection fraction <50%

Exclusion Criteria:

* Emergency surgery
* Withdrawal of consent
* Uncontrollable ventricular arrhythmias
* Obstructive cardiomyopathy
* Confirmed pregnancy test for women of child-bearing potential

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2005-05; Study Completion 2007-01 (Actual)

PRIMARY OUTCOMES:
pharmacokinetics | day of surgery

SECONDARY OUTCOMES:
hemodynamics | day of surgery

CONTACTS AND LOCATIONS:
Overall Officials: Jerrold H Levy, MD, Principal Investigator — Emory University
Locations (1):
- Emory University Hospital, Atlanta, Georgia, United States